CLINICAL TRIAL: NCT02678169
Title: A Prospective, Multicenter, Observational, Single-arm European Registry on the ACE Reperfusion Catheters and the Penumbra System in the Treatment of Acute Ischemic Stroke
Brief Title: European Registry on the ACE Reperfusion Catheters and the Penumbra System in the Treatment of Acute Ischemic Stroke
Acronym: PROMISE
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 9508
Record Dates: First submitted 2016-01-27; First posted 2016-02-09 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Penumbra Aspiration System: Penumbra Aspiration System with the ADAPT technique
  Interventions: Device: Penumbra Aspiration System

INTERVENTIONS:
Device: Penumbra Aspiration System — Penumbra Aspiration System using the ADAPT technique for recanalization of an occlusion large vessel in the brain

SUMMARY:
Prospective, single-arm, multicenter, observational registry of the ACE Reperfusion Catheters and the Penumbra System in Europe. Consecutive patients presenting within 6 hours from symptom onset with an acute ischemic stroke (within the internal carotid artery and internal carotid terminus, middle cerebral - M1/M2 segments) due to anterior circulation large vessel occlusion (LVO) will be treated using the ADAPT technique with thrombo-aspiration as first intention and site routine practice.

DETAILED DESCRIPTION:
Prospective, single-arm, multicenter, observational registry of the ACE Reperfusion Catheters and the Penumbra System in Europe. Consecutive patients presenting within 6 hours from symptom onset with an acute ischemic stroke (within the internal carotid artery and internal carotid terminus, middle cerebral - M1/M2 segments) due to anterior circulation large vessel occlusion (LVO) will be treated using the ADAPT technique with thrombo-aspiration as first intention and site routine practice.

The follow-up visit will occur 24 hours, 7-10 days or discharge, 30 days and 90 days post-procedure and will review patient's functional outcome, quality of life, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  * From 18 years of age
  * Present with symptoms consistent with an acute ischemic stroke within 6 hours of stroke symptom onset
  * Arterial occlusion of the distal intracranial carotid artery (ICA and ICA terminus) or middle cerebral artery (M1/M2)
  * National Institute of Health Stroke Scale (NIHSS) ≥ 2
  * Signed Informed Consent Form.

Imaging inclusion criteria:

• CT ASPECT score from 6 to 10 (>6) or according to MR DWI ASPECT score from 5 to 10 (>5).

Exclusion Criteria:

* General exclusion criteria:

  * Associated myocardial infarction or severe infection (endocarditis or sepsis)
  * Laboratory evidence of coagulation abnormalities, with an International Normalized Ratio (INR) of > 3.0 or platelets count < 40 x109/L or APTT > 50 sec
  * Uncontrolled hypertension (defined as systolic blood pressure > 185 mmHg or diastolic blood pressure > 110 mmHg)
  * Baseline glucose < 2.7 or > 22.2 mmol/L
  * Pre-stroke mRS score > 2
  * Seizure at the onset of stroke
  * Arterial tortuosity that would prevent the device from reaching the target vessel
  * Time of stroke symptoms onset unknown
  * Life expectancy less than 90 days prior to stroke onset
  * Females who are pregnant or lactating
  * Known serious sensitivity to radiographic contrast media.

Imaging exclusion criteria:

* CT/MRI evidence of the following conditions at screening:

  * Significant mass effect with midline shift
  * Evidence of intracranial hemorrhage (ICH), aneurysm, or arteriovenous malformation (AVM)
* Angiographic evidence of tandem extracranial occlusion or an arterial stenosis proximal to the occlusion that requires treatment prior to thrombus removal. Moderate stenosis not requiring treatment is not an exclusion criterion.
* Angiographic evidence of preexisting arterial injury, such as carotid dissection, complete cervical carotid occlusion, or vasculitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Present with symptoms consistent with an acute ischemic stroke within 6 hours of stroke symptom onset. Arterial occlusion of the distal intracranial carotid artery (ICA and ICA terminus) or middle cerebral artery (M1/M2)
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Angiographic revascularization of the occluded target vessel at immediate post-procedure as defined by a TICI 2b or 3 score. | Immediate post-procedure
Functional patient outcome at 90 days post-procedure as defined by a modified Rankin Score (mRS) 0-2. | 90 days post-procedure

SECONDARY OUTCOMES:
Incidence of device and procedure related Serious Adverse Events (SAEs) at 24 hours and 30 days from stroke treatment | 24 hours and 30 days from stroke treatment
All causes of mortality and morbidity at 90 days | 90 days
Occurrence of embolization in previously uninvolved (or new) territories (ENT) as seen on the final control angiogram at the end of procedure | At the end of interventional surgical procedure
Occurrence of symptomatic intracranial hemorrhages (sICH) at 24 hours | 24 hours
Occurrence of vessel damages at the end of the ADAPT procedure. | At the end of the interventional surgical procedure
NIHSS score at 7-10 days post-procedure. | 7-10 days post-procedure
Times to revascularization | From symptom onset to various times during the interventional surgical procedure
  * From symptom onset to CT-scan/MRI at the institution
  * From CT-scan/MRI at the institution to groin access
  * From groin puncture to final revascularization result.
Quality of Life: EQ-5D 3L score at 90 days compared to the one at 7-10 days post-procedure. | 90 days
Heath Economics: Total duration of hospitalization with related healthcare resources | Average time frame 3-7 days.
  * Health care professionals encountered/consulted before/after intervention
  * Tests performed before/after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schramm, MD, Principal Investigator — Universitätsklinikum Schleswig-Holstein, Lübeck, Germany
Locations (1):
- Universitätsklinikum Schleswig-Holstein, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schramm P, Navia P, Papa R, Zamarro J, Tomasello A, Weber W, Fiehler J, Michel P, Pereira VM, Krings T, Gralla J, Santalucia P, Pierot L, Lo TH. ADAPT technique with ACE68 and ACE64 reperfusion catheters in ischemic stroke treatment: results from the PROMISE study. J Neurointerv Surg. 2019 Mar;11(3):226-231. doi: 10.1136/neurintsurg-2018-014122. Epub 2018 Jul 30. PMID 30061367
- [Derived] Blanc R, Redjem H, Ciccio G, Smajda S, Desilles JP, Orng E, Taylor G, Drumez E, Fahed R, Labreuche J, Mazighi M, Lapergue B, Piotin M. Predictors of the Aspiration Component Success of a Direct Aspiration First Pass Technique (ADAPT) for the Endovascular Treatment of Stroke Reperfusion Strategy in Anterior Circulation Acute Stroke. Stroke. 2017 Jun;48(6):1588-1593. doi: 10.1161/STROKEAHA.116.016149. Epub 2017 Apr 20. PMID 28428348